CLINICAL TRIAL: NCT06655909
Title: Defining the Serum Ferritin Concentration in Kenyan Women and Their Preschool Children at Which the Body Senses Iron Depletion and Begins to Upregulate Iron Absorption From the Diet
Brief Title: Serum Ferritin Concentration in Kenyan Women and Their Preschool Children at Which the Body Begins to Upregulate Iron Absorption From the Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, PhD, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MOCHA
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer; Mothers; Preschool Children
Keywords: iron absorption; serum ferritin; maize porridge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mothers (Other): healthy volunteers
  Interventions: Other: consumption of maize porridge containing stable iron isotope
- preschool children (Other): healthy volunteers
  Interventions: Other: consumption of maize porridge containing stable iron isotope

INTERVENTIONS:
Other: consumption of maize porridge containing stable iron isotope — consumption of maize porridge containing stable iron isotope

SUMMARY:
Using standardized methods, the investigators will perform stable iron isotope absorption studies in young Kenyan women and their preschool children (2-5y of age) with varying iron status to measure iron absorption from maize meal containing labeled ferrous sulfate. Using these data, this study aim is to define the ferritin in these young women and children at which the body senses iron depletion and begins to upregulate iron absorption from the diet; this approach could provide a functionally defined threshold of iron deficiency in Sub-Saharan African women and children.

DETAILED DESCRIPTION:
In this experimental study in southern Kenya, the investigators will take a baseline venous blood sample to measure iron and inflammation biomarkers in generally healthy young women (n=125) and in their preschool children. The investigators will then administer, after an overnight fast, a standardized test meal porridge made from refined maize and bottled water containing the stable iron isotope 57Fe. Fourteen days later, the investigators will take a second venous blood sample for determination of erythrocyte incorporation of the 57Fe to measure iron absorption from the labeled test meal.

ELIGIBILITY:
Inclusion Criteria:

* < 75 kg
* BMI between 17 - 27.5 kg/m2
* No acute illness (self-reported)
* No metabolic or gastrointestinal disorders (self-reported)
* No use of medication affecting iron absorption or metabolism during the study
* No intake of mineral/vitamin supplements 2 weeks prior to the first study visit and during study
* Mother of a preschool age child (2-5 years)
* Child has normal Z-scores for WAZ, HAZ and WHZ (-3 - +3)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | Study day 14
  Erythrocyte iron incorporation

SECONDARY OUTCOMES:
Serum ferritin | Study day 1
  Serum ferritin concentration
soluble transferrin receptor | Study day 1
  soluble transferrin receptor concentration in serum
C-reactive protein | Study day 1
  C-reactive protein concentration in serum
alpha(1)-acid-glycoprotein | Study day 1
  alpha(1)-acid-glycoprotein concentration in serum

CONTACTS AND LOCATIONS:
Locations (1):
- ETH/JKUAT Research Station, Msambweni, Kenya

IPD SHARING:
Plan to Share IPD: No